CLINICAL TRIAL: NCT01834911
Title: Effect of Tetrabenazine on Stroop Interference in Huntington Disease
Brief Title: Effect of Tetrabenazine on Stroop Interference in HD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York Medical College (Other)
Responsible Party: Principal Investigator, Robert Fekete, Principal Investigator, New York Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L-10,830
Record Dates: First submitted 2013-04-15; First posted 2013-04-18 (Estimated); Results first posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Huntington Disease
Keywords: Huntington disease; HD; tetrabenazine; Stroop
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tetrabenazine withdrawal (Experimental): Tetrabenazine will be withdrawn for at least 3 days in Huntington disease patients currently taking the medication.
  Interventions: Drug: Tetrabenazine withdrawal

INTERVENTIONS:
Drug: Tetrabenazine withdrawal — Tetrabenazine will be withdrawn for at least 3 days in Huntington disease patients currently on the drug. Patients will be examined via Stroop test in the OFF state. Two doses of 12.5 mg tetrabenazine will be introduced, spaced 3 hours apart. Stroop test will be performed 6 hours after initial OFF Stroop test.

SUMMARY:
Tetrabenazine has been shown to improve gating of abnormal visual stimuli and improve postural stability in Huntington disease (HD) patients as measured by computerized dynamic posturography testing. This study aims to elucidate whether partial dopaminergic depletion via low dose tetrabenazine has a similar effect on masking out of abnormal visual stimuli on the Stroop interference test.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of Huntington disease by movement disorders expert
* Patients currently taking tetrabenazine.
* Patients should not have taken dopamine receptor blocking medication for at least three days

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Terence Cardinal Cooke Health Care Center, New York, New York, United States

REFERENCES:
- [Background] Fekete R, Davidson A, Ondo WG, Cohen HS. Effect of tetrabenazine on computerized dynamic posturography in Huntington disease patients. Parkinsonism Relat Disord. 2012 Aug;18(7):896-8. doi: 10.1016/j.parkreldis.2012.04.029. Epub 2012 May 22. PMID 22621818

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tetrabenazine Withdrawal
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tetrabenazine Withdrawal
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 57 [54 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Stroop Interference Score
Description: Participants will have Stroop Visual Interference Scores measured while OFF tetrabenazine for at least 3 days. Two doses of 12.5 mg tetrabenazine will be subsequently administered: first dose just after the Stroop test and second dose 3 hours later. Stroop Visual Interference Scores will be measured again in the ON state, 6 hours after the initial OFF measurement.
  Patients are analyzed according to Stroop test using Golden's Interference score (theoretical min -50, theoretical max about 98) calculated from [(W × C)/(W + C)] - CW, where C=color score (0-100), W=word score (0-100), CW=color word score (0-100). The Interference score analyzes cognitive interference during trials of reading of a list of color words which are printed in a different color. Lower or more negative scores are clinically better as they indicate less interference.
Time Frame: 72 hours
Population: Only 1 patient could complete all conditions of the Stroop test. The delta between on and off Stroop test was 1 using Golden's score [(W × C)/(W + C)] - CW
Measure: Number; unit: score on a scale
Arm/Group | Tetrabenazine Withdrawal
Number analyzed (Participants) | 1
score on a scale
  Interference score OFF | -1.97
  Interference score ON | -1

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Tetrabenazine Withdrawal
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Statistical analysis could not be performed as only one subject was able to provide complete study data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT01834911/Prot_SAP_000.pdf